CLINICAL TRIAL: NCT01201486
Title: Use of Color Doppler in Routine Examination of Fetal Heart in Second Trimester.
Status: Completed | Type: Observational
Sponsor: Helse Stavanger HF (Other Government)
Responsible Party: Sponsor
Other Study IDs: SUS-CH1
Record Dates: First submitted 2010-09-13; First posted 2010-09-14 (Estimated); Results first posted 2016-04-26 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Congenital Heart Defects
Keywords: Ultrasound; Pregnancy; Fetal heart defects; Color doppler
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pregnant women: Pregnant females in the 2nd trimester.

SUMMARY:
To evaluate the percentage of severe heart defect diagnosed with the use of color Doppler at a routine fetal scan in the second trimester of pregnancy

DETAILED DESCRIPTION:
Almost all women in Norway have a routine ultrasound examination in the second trimester, however, the detection rate of heart defect are only around 50%. In this study we use color Doppler at three different levels in the fetal heart; the four chamber view, the outlet of the aorta on on the level of the great arteries.

All heart defects at delivery are recorded and compared with the ultrasound findings.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* 2nd trimester

Exclusion Criteria:

* Unwilling

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women for routine examination in the 2nd trimester.
Sampling Method: Non-Probability Sample
Enrollment: 6781 (Actual)
Dates: Start 2006-10; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Heien, RN, Principal Investigator — Helse Stavanger HF; Torbjørn M. Eggebø, MD, Study Director — Helse Stavanger HF
Locations (1):
- Stavanger University Hospital, Stavanger, Norway

IPD SHARING:
Plan to Share IPD: No
Data wil not be shared outside the research group. Results are published (see references).

REFERENCES:
- [Background] Tegnander E, Eik-Nes SH, Johansen OJ, Linker DT. Prenatal detection of heart defects at the routine fetal examination at 18 weeks in a non-selected population. Ultrasound Obstet Gynecol. 1995 Jun;5(6):372-80. doi: 10.1046/j.1469-0705.1995.05060372.x. PMID 7552797
- [Background] Chaoui R, McEwing R. Three cross-sectional planes for fetal color Doppler echocardiography. Ultrasound Obstet Gynecol. 2003 Jan;21(1):81-93. doi: 10.1002/uog.5. PMID 12528169
- [Result] Eggebo TM, Heien C, Berget M, Ellingsen CL. Routine use of color Doppler in fetal heart scanning in a low-risk population. ISRN Obstet Gynecol. 2012;2012:496935. doi: 10.5402/2012/496935. Epub 2012 May 20. PMID 22685669

RESULTS

PARTICIPANT FLOW:
Groups:
- Pregnant Women in Second Trimester: Pregnant females in the 2nd trimester.
Period: Overall Study
Arm/Group | Pregnant Women in Second Trimester
Started | 6781
Completed | 6781
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The number of heart defects detected by color Doppler in the second trimester was compared to the number of major heart defects detected at birth to determine the sensitivity of the color Doppler examination to detect major heart defects in the second trimester.
Arm/Group | Pregnant Women in Second Trimester
Number analyzed (Participants) | 6781
Age, Continuous [Median (Full Range); unit: years] | 29 [16 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6781
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity of Color Doppler Examination to Detect Major Heart Defects During the Second Trimester of Pregnancy
Description: The number of *fetuses with* heart defects detected by color Doppler in the second trimester was compared to the number of *fetuses with* major heart defects detected at birth.
Time Frame: 2nd trimester
Measure: Number; unit: fetuses
Arm/Group | Pregnant Women
Number analyzed (Participants) | 6781
fetuses
  Major Heart Defects at Delivery | 39
  Heart Defects Detected by Color Dopple | 9
Statistical Analysis 1: Comparison: Pregnant Women; Test type: Superiority or Other; Percentage Sensitivity; Percentage Sensitivity = 23

ADVERSE EVENTS:
Arm/Group | Pregnant Women
Serious Adverse Events (participants affected / at risk) | 0/6781
Other Adverse Events (participants affected / at risk) | 0/6781

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes